CLINICAL TRIAL: NCT02501577
Title: Comparison of Various Supraglottic Airway Devices for Fiberoptical Guided Tracheal Intubation
Acronym: supraview
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Thomas Metterlein, MD, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: sadfoi
Record Dates: First submitted 2015-07-09; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Intubation; Difficult

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAD 1 (Experimental): FOI for placement
  Interventions: Device: SAD 1
- SAD 2 (Experimental): FOI für placement
  Interventions: Device: SAD 2

INTERVENTIONS:
Device: SAD 1 — Placement and fiberoptic control
  Arms: SAD 1
Device: SAD 2 — Placement and fiberoptic control
  Arms: SAD 2

SUMMARY:
Placement of a supraglottic airway device Fiberoptical verification of pharyngeal position

DETAILED DESCRIPTION:
Feasibility for fiberoptical verification of pharyngeal position of supraglottic airway device

ELIGIBILITY:
Inclusion Criteria:

* will to participate

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Visibility of vocal cords | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Metterlein, MD, Study Chair — Uni Regensburg
Locations (1):
- University Regensburg, Regensburg, Germany